CLINICAL TRIAL: NCT05550363
Title: A Phase 3, Prospective, Randomized, Double-masked, Placebo-controlled, Parallel-design, Multicenter Study to Evaluate the Efficacy and Safety of DEXYCU® for the Treatment of Ocular Pain Associated With Cataract Surgery
Brief Title: A Study to Evaluate the Efficacy and Safety of DEXYCU® for the Treatment of Ocular Pain Associated With Cataract Surgery (2)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Not currently pursuing indication
Sponsor: EyePoint Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EYP-DIP-302
Record Dates: First submitted 2022-09-16; First posted 2022-09-22 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2022-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Double-masked, Placebo-controlled,Parallel-design, Multicenter Study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DEXYCU (Experimental): DEXYCU, 103.4 mcg/mcl dexamethasone: equivalent dexamethasone dose: 517 mcg
  Interventions: Drug: Dexycu
- Placebo (Placebo Comparator): Placebo/vehicle, 0 mcg/mcl dexamethasone: equivalent dexamethasone dose: 0 mcg
  Interventions: Other: Placebo/Vehicle

INTERVENTIONS:
Drug: Dexycu — 103.4 mcg/mcl dexamethasone: equivalent dexamethasone dose: 517 mcg
  Arms: DEXYCU
Other: Placebo/Vehicle — Placebo/vehicle, 0 mcg/mcl dexamethasone: equivalent dexamethasone dose: 0 mcg
  Arms: Placebo

SUMMARY:
A Phase 3, Prospective, Randomized, Double-masked, Placebo-controlled, Parallel-design, Multicenter Study to Evaluate the Efficacy and Safety of DEXYCU® for the Treatment of Ocular Pain Associated with Cataract Surgery

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 40 years of age scheduled for cataract surgery
* Best corrected visual acuity (BCVA) of 20/30-20/200 in the study eye
* Must be considered by the investigator to have visual (VA) acuity potential greater than 20/30 in the study eye.

Exclusion Criteria:

* Use of any corticosteroids within 7 days prior to Day 0
* Injection of any corticosteroids, systemic immunomodulators or alkylating agents into any body tissue within 90 days
* Score greater than "0" on the Ocular Pain Assessment in the study eye at Screening.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with absence of ocular pain (ie, score of '0') in the study eye at Day 8 | Day 8

SECONDARY OUTCOMES:
Proportion of subjects with absence of ocular pain in the study eye at Days 1, 3, 15, and 30 | Days 1, 3, 15, and 30
Mean ocular pain scores in the study eye | Days 1, 3, 15, and 30
  Numerical Ocular Pain Scale from 0-10 with 0 being no pain and 10 being most severe
Proportion of subjects with absence of cells in the AC of the study eye | Days 1, 3, 15, and 30
Proportion of subjects with absence of flare in the AC of the study eye | Days 1, 3, 15, and 30
Mean AC cell score in the study eye | Days 1, 3, 15, and 30
  AC count by Slit Lamp Biomicroscopy with 0 being none and 4 being most severe
Mean AC flare score in the study eye | Days 1, 3, 15, and 30
  AC flare by Slit Lamp Biomicroscopy with 0 being absent and 4 being strong intensity
Rates of ocular (study eye and fellow eye) and non-ocular TEAEs | up to day 30

IPD SHARING:
Plan to Share IPD: No